CLINICAL TRIAL: NCT00267735
Title: Measuring Preferences for Childbirth After Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1R03HS013959-01A1 (AHRQ)
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Pregnancy
Keywords: pregnancy; repeat cesarean; vaginal birth after cesarean

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Module 1 Only (No Intervention)
- Modules 1, 2, and 3 (Experimental)
  Interventions: Behavioral: Use of Computerized Decision Aid on Childbirth

INTERVENTIONS:
Behavioral: Use of Computerized Decision Aid on Childbirth
  Arms: Modules 1, 2, and 3

SUMMARY:
The objective of this proposed 18-month exploratory research study is to help pregnant women weigh risks and benefits in a childbirth decision using the Preferences-Assessment Computer Module. Our hypothesis is that, after using this computer module, women will be more aware of the potential risks and benefits of VBAC and of elective repeat cesarean and will have greater clarity about their preferences related to these risks and benefits.

DETAILED DESCRIPTION:
As cesarean birth rates continue to climb, the number of women (currently about 420,000 annually) facing the decision of whether to have a repeat cesarean or to attempt a vaginal birth after cesarean (VBAC) will also increase. The objective of this proposed 18-month exploratory research study is to help pregnant women weigh risks and benefits in a childbirth decision using the Preferences Assessment Computer Module developed by the principal investigator. The long-term objective of the proposed research is to understand and improve the decision-making process of these women by creating a computerized childbirth decision aid. Such decision aids provide value when the decision is complex, when the outcome is uncertain, and when people vary in how they prioritize preferences; childbirth decisions for women with a prior cesarean meet all these criteria.

No study to date quantifies how women weigh the complexities of various considerations-medical and otherwise-in the delivery decision. The proposed research is significant, therefore, in that it will provide a much-needed method to help women prioritize and weigh their preferences related to childbirth decisions. More broadly, it responds to the recent NIH and AHRQ initiatives to promote the development of computerized decision aids to improve the quality of medical decisions.

A new investigator will lead a well-qualified, multi-disciplined team that has expertise in decision analysis, obstetric medicine, and research methodology in pursuit of the following specific aims:

1. To validate a precise method to measure childbirth preferences. During the initial phase of this study, we will verify the accuracy of the Preferences Assessment Computer Module, measure internal consistency and assess content validity in a cross-sectional study.
2. To test whether women who use the Preferences Assessment Computer Module will have increased clarity about their preferences-and about the implication of those preferences-in comparison to women in a control group. We will conduct a randomized controlled trial of pregnant women with a prior cesarean.

This Preferences Assessment Computer Module is appropriate to address not only VBAC decisions, but also decisions related to elective cesareans and induction. In short, the proposed research will advance the field by improving the quality of the decision-making process for childbirth.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* pregnant
* candidate for VBAC
* singleton pregnancy
* one prior cesarean
* with a non-vertical uterine scar
* English or Spanish speaking

Exclusion Criteria:

* more than one prior cesarean

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Decisional conflict scores (knowledge of options; clarity about preferences; decisional certainty; conflict) after using decision aid.

CONTACTS AND LOCATIONS:
Overall Officials: Karen B Eden, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University Clinics, Portland, Oregon, United States